CLINICAL TRIAL: NCT03578744
Title: Efficacy of Platelet Rich Fibrin as a Graft and Membrane Versus Hyaluronic Acid and Amniotic Membrane in the Treatment of Mandibular Grade II and Grade III Furcation Defects- A Randomized Clinical Trial
Brief Title: Comparison of Platelet Rich Fibrin as Graft & Membrane Vs Hyaluronic Acid & Amniotic Membrane in the Treatment of Interradicular Defects
Acronym: CPRFGMHATID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Boyeena Lavanya, Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMIDS; 16201105031D (Other: Kaloji Narayana Rao University of Health Sciences.)
Record Dates: First submitted 2018-05-31; First posted 2018-07-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Intervention Model Description: Patients will be equally divided into two test groups, Group A and Group B after phase I therapy. The group A patients will be treated with conventional flap surgery and the furcation would be debrided, following which platelet-rich fibrin will be placed as a graft and a membrane. The flap will then be sutured back. The group B patients will also be treated with conventional flap surgery after furcation area is debrided, and hyaluronic acid (gengigel)will be placed as a graft over which amniotic membrane will be placed. The flap would then be sutured.
Who Masked: Participant
Masking Description: Sealed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Group A patients will be treated with conventional flap surgery. The furcation defects will be debrided and autologous platelet-rich fibrin will be paced as a graft and membrane. Later the flap will be sutured.
  Interventions: Procedure: Conventional Flap surgery
- Interventional Comparator (Experimental): Group B patients will be treated with conventional flap surgery. The furcation defects will be debrided and Hyaluronic acid (Gengigel) will be placed as a graft. Amniotic membrane (Tata Memorial Hospital Mumbai) will be placed over the graft and later the flap will be sutured.
  Interventions: Procedure: Conventional Flap surgery

INTERVENTIONS:
Procedure: Conventional Flap surgery — After administering local anaesthetic a full thickness flap will be raised and reflected to expose the furcation defects. The furcation defects would then be debrided and the graft and membrane secured in position. Later the flap would be sutured back.

SUMMARY:
This study is intended to compare the efficacy of platelet-rich fibrin as a graft and a membrane versus hyaluronic acid(Gengigel) and amniotic membrane in the treatment of mandibular grade II furcation defects.

DETAILED DESCRIPTION:
Platelet-rich fibrin is a fraction of plasma that provides a rich source of growth factors and may enhance the stabilization and revascularization of the flaps and grafts.

Hyaluronic acid is a naturally occurring non-sulfated high molecular weight glycosaminoglycan that forms a critical component of the extracellular matrix and contributes significantly to tissue hydrodynamics, cell migration and proliferation. Hence its administration to periodontal wound sites could achieve beneficial effects in periodontal tissue regeneration.

Amniotic membrane is being used for various regenerative procedures as it is a rich source of various collagen and non-collagen proteins such as laminin, fibronectin and proteoglycan.

ELIGIBILITY:
Inclusion Criteria:

* Grade II furcation involvement

Exclusion Criteria:

* Smokers,
* Pregnant and lactating women,
* Systemically compromised patients

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Radiological Parameters | Baseline and 9 months post surgery.
  Amount of Bone fill in the furcation (Change in Bone level) to be measured by Cone Beam Computed Tomography(CBCT)

SECONDARY OUTCOMES:
Clinical Parameter | Baseline and 9 months post surgery.
  Change in relative vertical clinical attachment level will be measured by Williams probe in millimeters in the furcation area.
Clinical Parameter | Baseline and 9 months post surgery
  Change in relative horizontal clinical attachment level will be measured in millimeters by the Nabers probe in the furcation area

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Boyeena, (MDS), Principal Investigator — PG Student
Locations (1):
- Dr.Rekha Rani Koduganti, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kothiwale SV, Anuroopa P, Gajiwala AL. A clinical and radiological evaluation of DFDBA with amniotic membrane versus bovine derived xenograft with amniotic membrane in human periodontal grade II furcation defects. Cell Tissue Bank. 2009 Nov;10(4):317-26. doi: 10.1007/s10561-009-9126-3. Epub 2009 Mar 10. PMID 19277899
- [Background] Sharma A, Pradeep AR. Autologous platelet-rich fibrin in the treatment of mandibular degree II furcation defects: a randomized clinical trial. J Periodontol. 2011 Oct;82(10):1396-403. doi: 10.1902/jop.2011.100731. Epub 2011 Feb 2. PMID 21284545